CLINICAL TRIAL: NCT06658080
Title: Drug Sensitivity Based on Hydrothorax and Ascite Organoids Derived from Metastasic Breast Cancer
Brief Title: Drug Sensitivity of Hydrothorax and Ascite Organoids from Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0866
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer Metastatic; Hydrothorax; Ascites; Organoids; Drug Evaluation
MeSH Terms: conditions — Hydrothorax; Ascites

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: organoid drug test — Before initiating therapy, patients diagnosed with metastatic breast cancer patients with hydrothorax and ascite fluid. The hydrothorax and ascite fluid is utilized to establish organoids and conduct drug testing.

SUMMARY:
Malignant hydrothorax and ascitic fluid in advanced breast cancer often arise from metastasis to the lungs, pleura, or liver. Patients with this condition experience rapid disease progression and multidrug resistance, facing limited treatment options. Clinical guidelines offer various therapies based on molecular subtypes; however, their effectiveness can be hindered by prior treatments, patient health, and tumor evolution. Current evaluations of treatment efficacy typically take two cycles, delaying the recognition of ineffective therapies and resulting in unnecessary side effects and costs. Organoid models present a promising solution, accurately replicating tumor structure and cellular diversity compared to traditional methods. These patient-derived models facilitate improved drug sensitivity testing, leading to more personalized treatment plans. In this study, 90 patients diagnosed with metastatic breast cancer accompanied by hydrothorax and ascitic fluid will be recruited. Patient-derived organoids will be used to assess the sensitivity of chemotherapy regimens, including Doxorubicin, Carboplatin, Cyclophosphamide, and Paclitaxel, along with targeted therapies such as Herceptin and Pertuzumab.

DETAILED DESCRIPTION:
90 metastatic breast cancer patients with hydrothorax and ascitic fluid will be recruited. Baseline data, including medical history, ultrasound, and MRI records, will be collected both before and after two cycles of chemotherapy. Tumor samples from hydrothorax and ascitic fluid will be obtained and cultured to generate patient-derived organoids (PDOs). These PDOs will then be exposed to standard chemotherapeutic drugs used in breast cancer treatment. Organoid growth will be monitored post-treatment, and dose-response curves will be generated to assess drug sensitivity. To evaluate clinical outcomes, the RECIST criteria will be applied to measure tumor response in patients. Correlation analysis will be performed to determine the consistency between the treatment responses observed in the PDO models and the actual clinical outcomes of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form and willingness to participate in the clinical study.
2. patients aged between 18 and 70 years old.
3. Confirmed metastatic breast cancer patients with hydrothorax and ascite fluid, which was verified to contain tumor cells by lab.
4. ECOG performance status score of 0-1.
5. No significant abnormalities in liver and kidney function (BIL <1.5-fold upper limit of normal (ULN)；ALT<2.5×ULN; AST<2.5×ULN；Crea≤1×ULN).

Exclusion Criteria:

1.Patients not suitable for chemotherapy and target therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: metastatic breast cancer patients with hydrothorax and ascite fluid
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-11-09 (Actual); Primary Completion 2026-10-25 (Estimated); Study Completion 2027-10-25 (Estimated)

PRIMARY OUTCOMES:
Correlation between drug sensitivity test results in patient-derived organoid models and clinical outcomes. The drug sensitivity test results obtained from patient-derived organoid models will be compared with the clinical outcomes. | 2024.10-2026.10

SECONDARY OUTCOMES:
The sensitivity and specificity would be checked between drug sensitivity of organoid models in predicting the efficacy of treatment. | 2024.10-2026.10

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Second affiliated hospital of zhejiang university, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - 2 nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No